CLINICAL TRIAL: NCT02440022
Title: A Prospective, Global, Multicenter, Randomized, Controlled Study Comparing Lutonix® 035 AV Drug Coated Balloon PTA Catheter vs. Standard Balloon PTA Catheter for the Treatment of Dysfunctional AV Fistulae
Brief Title: Study Comparing Lutonix AV Drug Coated Balloon vs Standard Balloon for Treatment of Dysfunctional AV Fistulae
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL0023-01
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lutonix DCB (Experimental): Percutaneous transluminal angiography (PTA) will be performed using the Lutonix AV drug coated balloon.
  Interventions: Combination Product: Lutonix DCB; Procedure: Percutaneous Transluminal Angiography
- Standard Balloon Angioplasty Catheter (Active Comparator): Percutaneous transluminal angiography (PTA) will be performed using a commercially available uncoated PTA balloon. Balloons with an external wire support, cutting/scoring component or other similar modifications are not permitted. Multiple balloons, inflations and/or prolonged inflation may be used.
  Interventions: Device: Standard Balloon Angioplasty Catheter; Procedure: Percutaneous Transluminal Angiography

INTERVENTIONS:
Combination Product: Lutonix DCB
  Arms: Lutonix DCB
Device: Standard Balloon Angioplasty Catheter
  Arms: Standard Balloon Angioplasty Catheter
Procedure: Percutaneous Transluminal Angiography — Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
  Other Names: PTA

SUMMARY:
This prospective, global, multicenter, randomized, controlled study is designed to evaluate the safety and effectiveness of the Lutonix 035 AV Drug Coated Balloon PTA Catheter compared to a standard PTA Catheter in treating subjects presenting with clinical and hemodynamic abnormalities in native arteriovenous (AV) fistulae located in the upper extremity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years;
2. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form (ICF);
3. Arteriovenous fistula located in the arm;
4. Native AV fistula was created ≥30 days prior to the index procedure and has undergone one or more hemodialysis sessions;
5. Venous stenosis of an AV fistula with the target lesion located from the anastomosis to the axillosubclavian junction and an abnormality attributable to the stenosis as defined by K/DOQI guidelines.;
6. Successful pre-dilation of the target lesion with a percutaneous transluminal angioplasty (PTA) balloon;
7. Intended target lesion.

Exclusion Criteria:

1. Women who are pregnant, lactating, or planning on becoming pregnant during the study;
2. Hemodialysis access is located in the leg;
3. Subject has more than two lesions in the access circuit;
4. Subject has a secondary non-target lesion that cannot be successfully treated;
5. Target lesion is located central to the axillosubclavian junction;
6. The subject has a secondary lesion located in the central venous system (central to the axillosubclavian junction);
7. A thrombosed access;
8. Surgical revision of the access site planned;
9. Recent prior surgical interventions of the access site;
10. Other planned treatment during the index procedure;
11. Known contraindication (including allergic reaction) or sensitivity to iodinated contrast media, that cannot be adequately managed with pre-and post-procedure medication;
12. Known contraindication (including allergic reaction) or sensitivity to paclitaxel.
13. Subjects who are taking immunosuppressive therapy or are routinely taking

    ≥10mg of prednisone per day;
14. Subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be noncompliant with the protocol or confound the data interpretation;
15. Subject has a life expectancy <12 months;
16. Anticipated for a kidney transplant;
17. Anticipated conversion to peritoneal dialysis;
18. Subject has a stent located in the target or secondary non target lesion;
19. Subject has an infected AV access or systemic infection;
20. Currently participating in an investigational drug, biologic, or device study, or previous enrollment in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Trerotola, MD, Principal Investigator — University of Pennsylvania
Locations (23):
- United States (23):
  - The Board of Trustees of The University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Kidney Disease and Hypertension Center Medical Research Services, LLC, Phoenix, Arizona
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - Capital Nephrology Medical Group, Sacramento, California
  - Nephrology Associates, P.A., Newark, Delaware
  - Rush University, Chicago, Illinois
  - RenalCare Associates, S.C. d/b/a Illinois Kidney Disease & Hypertension Center, Peoria, Illinois
  - MakrisMD, LLC, d/b/a Chicago Access Care, Westmont, Illinois
  - Massachusetts General Physicians Organizations, Inc., Boston, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - Michigan Vascular Center, Flint, Michigan
  - Minnesota Vascular Surgery Center, New Brighton, Minnesota
  - Capital Nephrology Associates, P.A., Raleigh, North Carolina
  - Oklahoma Life Access, PLLC, Tulsa, Oklahoma
  - Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Providence Interventional Associates, LLC, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Regional Health Services District, Inc., Spartanburg, South Carolina
  - University Vascular Access, Memphis, Tennessee
  - Tarrant Vascular Clinic, Fort Worth, Texas
  - San Antonio Kidney Disease Center Physicians Group, PLLC, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Board of Regents of the University of Wisconsin System, Madison, Wisconsin

REFERENCES:
- [Derived] Trerotola SO, Lawson J, Roy-Chaudhury P, Saad TF; Lutonix AV Clinical Trial Investigators. Drug Coated Balloon Angioplasty in Failing AV Fistulas: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2018 Aug 7;13(8):1215-1224. doi: 10.2215/CJN.14231217. Epub 2018 Jul 24. PMID 30042225

RESULTS

PARTICIPANT FLOW:
Groups:
- Lutonix DCB: Percutaneous transluminal angiography (PTA) will be performed using the Lutonix AV drug coated balloon.
  Lutonix DCB
  Percutaneous Transluminal Angiography: Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
- Standard Balloon Angioplasty Catheter: Percutaneous transluminal angiography (PTA) will be performed using a commercially available uncoated PTA balloon. Balloons with an external wire support, cutting/scoring component or other similar modifications are not permitted. Multiple balloons, inflations and/or prolonged inflation may be used.
  Standard Balloon Angioplasty Catheter
  Percutaneous Transluminal Angiography: Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
Period: Overall Study
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Started | 141 | 144
Completed | 114 | 131
Not Completed | 27 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter | Total
Number analyzed (Participants) | 141 | 144 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (14.46) | 61 (13.36) | 62.3 (13.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 59 | 113
  Male | 87 | 85 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 28 | 49
  Not Hispanic or Latino | 120 | 116 | 236
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 141 | 144 | 285

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Primary Patency (TLPP) at 6 Months Post Index Procedure
Description: Primary Patency is defined as the interval following index procedure intervention until clinically driven reintervention of the target lesion or access thrombosis. Target Lesion Primary Patency (TLPP) ends with a clinically driven re-intervention of the target lesion or access thrombosis.
Time Frame: 6 months post index procedure
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Percentage of Participants | 71.4 [62.7 to 78.4] | 63 [54.4 to 70.4]
Statistical Analysis 1: Comparison: Lutonix DCB vs Standard Balloon Angioplasty Catheter; Test type: Superiority; p = 0.0562, Kaplan-Meier

2. Primary Outcome: Number of Participants With Freedom From Any Serious Adverse Event(s) Involving the AV Access Circuit at 30 Days Post Index Procedure.
Description: The primary safety endpoint is freedom from localized or systemic serious adverse events through 30 days that reasonably suggests the involvement of the AV access circuit (CEC adjudicated).
Time Frame: 30 Days Post Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 137 | 144
Participants | 130 | 138
Statistical Analysis 1: Comparison: Lutonix DCB vs Standard Balloon Angioplasty Catheter; H0: The primary safety rate p1 in the DCB treatment group through 30 days post index procedure is inferior to that p2 of the PTA treatment group. (i.e. p1 ≤ p2 - δ) H1: The primary safety rate p1 in the DCB treatment group through 30 days post index procedure is non-inferior to that p2 of the PTA treatment group. (i.e. p1 > p2 - δ); Test type: Non-Inferiority — Where δ = 10% is the non-inferiority margin, which is the range of difference that is considered not clinically important. A non-inferiority Farrington and Manning Test was used to test the primary safety hypothesis. The test is successful if the one-sided p-value is less than 0.025. In addition to the p-value of the test, the confidence intervals of the rate in each group and the difference between the two groups is calculated; p = 0.002, Binary Analysis

3. Secondary Outcome: Percentage of Participants With Target Lesion Primary Patency at 3, 9, 12, 18, and 24 Months
Description: as for outcome 1
Time Frame: 3, 9, 12, 18, and 24 Months Post Index Procedure
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Percentage of Participants
  At 3 months | 92.6 [86.6 to 95.9] | 86.7 [79.9 to 91.3]
  At 9 months | 58 [48.8 to 66.1] | 46.4 [37.8 to 54.5]
  At 12 months | 44.4 [35.3 to 53.1] | 36 [27.9 to 44.2]
  At 18 months | 34 [25.3 to 42.9] | 28.3 [20.8 to 36.3]
  At 24 months | 26.9 [18.6 to 35.8] | 24.4 [17.2 to 32.3]

4. Secondary Outcome: Percentage of Participants With Device, Procedural and Clinical Success
Description: * Device Success: Successful delivery to the target lesion, deployment, and retrieval at index procedure.
  * Procedural Success: At least one indicator of hemodynamic success (e.g., physical examination with restoration of a thrill, direct measurement of flow) in the absence of peri-procedural (index procedure and through hospital stay) Serious Adverse Device Effects (SADEs).
  * Clinical Success: The resumption of dialysis for at least one session after the index procedure.
Time Frame: Device and Procedural Success: At time of Index Procedure; Clinical Success: at 1st session of dialysis following index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Percentage of participants
  Device Success | 100 | 100
  Procedure Success | 97.9 | 99.3
  Clinical Success | 99.3 | 100

5. Secondary Outcome: Number of Participants With Abandonment of Permanent Access in the Index Extremity at 3, 6, 9, 12, 18, and 24 Months Post Index Procedure
Description: Index access site abandonment refers to an abandonment due to either receiving a kidney transplant, converting to Peritoneal Dialysis, or a new access site being created.
Time Frame: 3, 6, 9, 12, 18 and 24 Months Post Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Participants
  At 3 months | 3 | 0
  At 6 months | 5 | 1
  At 9 months | 12 | 4
  At 12 months | 13 | 6
  At 18 months | 14 | 10
  At 24 months | 22 | 13

6. Secondary Outcome: Number of Interventions Required to Maintain Access Circuit Primary Patency (ACPP) at 3, 6, 9, 12, 18, and 24 Months Post Index Procedure
Time Frame: 3, 6, 9, 12, 18 and 24 Months Post Index Procedure
Measure: Number; unit: Interventions
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Interventions
  At 3 months | 21 | 20
  At 6 months | 68 | 78
  At 9 months | 115 | 126
  At 12 months | 164 | 181
  At 18 months | 228 | 252
  At 24 months | 291 | 321

7. Secondary Outcome: Number of Participants With Device Related Adverse Events at 1, 3, 6, 9, 12, 18, and 24 Months (CEC Adjudicated)
Description: Events adjudicated as 'definitely related' and 'possibly related' by the CEC were combined in all analyses and are displayed as 'related' in this report.
Time Frame: 1, 3, 6, 9, 12, 18 and 24 Months Post Index Procedure
Population: CEC adjudicated.
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Participants
  At 1 month | 5 | 1
  At 3 months | 7 | 2
  At 6 months | 7 | 2
  At 9 months | 7 | 2
  At 12 months | 7 | 2
  At 18 months | 7 | 2
  At 24 months | 7 | 2

8. Secondary Outcome: Number of Participants With Target Lesion Primary Patency (TLPP) by Fiber Pre-Dilation Balloon at 6 Months Post Index Procedure
Description: as for outcome 1
Time Frame: 6 Months Post Index Procedure
Population: The (n) analyzed depended on the number of participants for which data was available at the time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Participants
  Fiber: number analyzed (Participants) | 82 | 80
  Fiber | 57 | 48
  Non-Fiber: number analyzed (Participants) | 44 | 59
  Non-Fiber | 32 | 40
Statistical Analysis 1: Comparison: Lutonix DCB vs Standard Balloon Angioplasty Catheter; Test type: Other; p = 0.7160, Regression, Cox — P-value was type 3 test of the interaction of treatment group and pre-dilation balloon type

9. Secondary Outcome: Number of Interventions Required to Maintain Target Lesion Primary Patency (TLPP) at 3, 6, 9, 12, 18, and 24 Months Post Index Procedure
Time Frame: 3, 6, 9, 12, 18, and 24 Months Post Index Procedure
Measure: Number; unit: Interventions
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Interventions
  At 3 months | 19 | 11
  At 6 months | 44 | 64
  At 9 months | 66 | 93
  At 12 months | 113 | 137
  At 18 months | 160 | 184
  At 24 months | 208 | 223

10. Secondary Outcome: Number of Procedure Related Serious Adverse Events (CEC Adjudicated) at 1, 3, 6, 9, 12, 18, and 24 Months Post Index Procedure
Time Frame: 1, 3, 6, 9, 12, 18, and 24 Months Post Index Procedure
Measure: Number; unit: Events
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 141 | 144
Events
  At 1 month | 8 | 2
  At 3 Months | 11 | 3
  At 6 Months | 11 | 4
  At 9 Months | 11 | 4
  At 12 Months | 11 | 4
  At 18 Months | 11 | 4
  At 24 Months | 11 | 4

ADVERSE EVENTS:
Time Frame: At 24 months Post Index Procedure
Description: The Serious Adverse Events (SAEs) presented reflect Subjects with SAEs by body system and preferred term (CEC adjudicated) at 24 months post index procedure.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
All-Cause Mortality (participants affected / at risk) | 33/141 | 26/144
Serious Adverse Events (participants affected / at risk) | 115/141 | 123/144
Other Adverse Events (participants affected / at risk) | 97/141 | 114/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix DCB (N=141) | Standard Balloon Angioplasty Catheter (N=144)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 6 | 6
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 3
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Cardiac death (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 6 | 6
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 94 | 110
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 13 | 17
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Injury (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 7 | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Brachiocephalic vein stenosis (Vascular disorders) | 2 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Steal syndrome (Vascular disorders) | 2 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Venous occlusion (Vascular disorders) | 9 | 14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix DCB (N=141) | Standard Balloon Angioplasty Catheter (N=144)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 94 (94) | 110 (110)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 13 (13) | 17 (17)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Brachiocephalic vein stenosis (Vascular disorders) | 2 (2) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 1 (1) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular calcification (Vascular disorders) | 0 (0) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Venous occlusion (Vascular disorders) | 9 (9) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT02440022/Prot_SAP_000.pdf